CLINICAL TRIAL: NCT06980532
Title: Glumetinib Combined With Fruquintinib in the Treatment of MET Amplification or Protein Overexpression in Third-Line Unresectable Metastatic Colorectal Cancer: A Prospective, Exploratory, Open-Label Clinical Study
Brief Title: Glumetinib Combined With Fruquintinib in the Treatment of MET Amplification or Protein Overexpression in Third-Line Unresectable Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liu Huang (Other)
Responsible Party: Sponsor-Investigator, Liu Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202502131
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glumetinib combined with Fruquintinib (Experimental)
  Interventions: Drug: Glumetinib Combined with Fruquintinib

INTERVENTIONS:
Drug: Glumetinib Combined with Fruquintinib — Fruquintinib: 3mg, po.qd, d1-14，q3w;
  Guemitinib:
  Grade 1:200mg, po, qd, q3w; Grade 2:250mg, po, qd, q3w; Phase I: The dose of Glumetinib (200 mg → 250 mg) is dynamically adjusted using the "3+3 dose-escalation rule" to determine the optimal dose of Fruquintinib.
  Phase II: The RP2D (Recommended Phase II Dose) of Glumetinib identified in Phase I is continued in combination with Fruquintinib.

SUMMARY:
Glumetinib combined withFruquintinib in the treatment of MET amplification or protein overexpression in third-line unresectable metastatic colorectal cancer: evaluation of efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. The patients fully understood this study, voluntarily participated and signed the Informed Consent Form (ICF);
2. Age ≥18 years old;
3. Patients with unresectable metastatic colorectal cancer with microsatellite stable (MSS) confirmed by pathology or histology;
4. Have MET amplification (FISH MET GCN≥4 or MET/CEP7≥1.8; Or NGS, ≥20% of tumor cells, ≥200X sequencing depth, GCN≥4) or overexpression (IHC, 3+(≥50% of tumor cells are strongly positive) or 2+ (≥50% of tumor cells are moderately positive/strongly positive and < 50% of tumor cells are strongly positive); Immunohistochemistry (IHC) detection showed that the MET protein overexpression in the subjects was 3+(strongly positive in ≥50% of tumor cells) or 2+ (positive in ≥50% of tumor cells/weakly positive and strongly positive in < 50% of tumor cells).
5. Imaging confirmed progression after previous two-line standard anti-tumor regimens;
6. According to RECIST1.1 criteria, the patient has at least one measurable target lesion; For lesions that have undergone radiotherapy in the past, they can only be included in measurable lesions when there is clear disease progression after radiotherapy.
7. Eastern Cooperative Oncology Group (ECOG) Physical Status Score: 0-1 point;
8. The expected survival time is ≥3 months;
9. Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥75×10^9/L and hemoglobin 80 g/L, white blood cell count (WBC) ≥3.0×10^9/L (corrected by no blood transfusion, no blood products, no use of granulocyte colony-stimulating factor or other hematopoietic stimulating factor within 14 days before laboratory tests);
10. Liver and kidney functions: Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance rate ≥50mL/min; AST and ALT ≤2.5 times the upper limit of normal values (for patients with liver invasion, ≤5 times the upper limit of normal values); Serum total bilirubin ≤2 times the upper limit of normal value (for patients with liver invasion ≤2.5 times the upper limit of normal value);
11. The activated partial thromboplastin time (APTT), International normalized ratio (INR), and prothrombin time (PT) are ≤1.5 times the normal upper limit value.
12. Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, with a negative result, and be willing to use appropriate contraceptive methods (such as intrauterine devices [IUD], contraceptives or condoms) during the test and 6 months after the last administration of the test drug; The serum pregnancy test must be negative within 7 days before enrollment in the study, and the subjects must be non-lactating. Male subjects who should agree that contraceptive measures must be adopted during the study period and within 6 months after the end of the study period;

Exclusion Criteria:

Have received MET inhibitor treatment in the past; 2. Patients with unresectable metastatic colorectal cancer who have MSI-H/dMMR (MSI detection shows instability at two or more sites, and MMR detection shows loss of expression at any one protein); 3. Patients with unresectable metastatic colorectal cancer whose BRAF gene test is mutant and who have not received BRAF inhibitors /MEK inhibitors; 4. Patients with severe active bleeding, active peptic ulcers, unhealed gastrointestinal perforations, and peptic fistulas; 5. Have hypersensitivity reactions to any investigational drug or its components; 6. Concurrent severe and uncontrolled concurrent infections or other severe and uncontrolled concomitant diseases, moderate or severe renal injury; (such as progressive infection, uncontrollable hypertension, diabetes, etc.) 7. Infection during the active stage of hepatitis B and C (positive hepatitis B virus surface antigen and hepatitis B virus DNA exceeding 1 × 103 copies /mL; Hepatitis C virus RNA exceeds 1 × 103 copies /mL; 8. Human immunodeficiency virus (HIV) infection (HIV antibody positive); 9. Have had or are currently suffering from other malignant tumors simultaneously (except for effectively controlled non-melanoma basal cell carcinoma of the skin, breast/cervical carcinoma in situ, and other malignant tumors that have been effectively controlled without treatment in the past five years); 10. Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures; 11. Those with other malignant tumors requiring treatment; 12. The researchers judged that patients were not suitable to participate in this study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended dose for Phase II | Up to approximately 18 Weeks
  The dose determined during dose-escalation trials for use in Phase II studies, typically based on safety and tolerability data.
Objective response rate(ORR) | Up to approximately 18 Weeks
  In the phase II study,CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Maximum tolerated dose(MTD) | Up to approximately 18 Weeks
  The highest dose identified in dose-escalation trials that does not cause dose-limiting toxicities (DLTs).
Dose-limiting toxicity（DLT） | Up to approximately 18 Weeks
  Severe or intolerable toxicity events related to the study drug within a specified time window, which may influence dose-escalation decisions.
Assess Adverse Events | up to 12 months
  Assess adverse events according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Disease control rate（DCR） | Up to approximately 18 Weeks
  Proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD).
Overall Survival (OS) | Up to approximately 36 Months
  Overall survival is defined as the time from enrollment to death due to any cause.
Objective Response Rate (ORR) | Up to approximately 18 Weeks
  In Phase I studies, CR + PR rate according to the RECIST version 1.1 guidelines.
Progression-free survival（PFS） | Up to approximately 18 Weeks
  Time from enrollment to disease progression (based on imaging or clinical assessment) or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No